CLINICAL TRIAL: NCT01794949
Title: Optical Frequency Domain Imaging (OFDI) Determined Stent Strut Coverage and Plaque Morphology After RESOLUTE Stent Placement in Non-Insulin Dependent Diabetics Presenting With Acute Coronary Syndrome (ACS)
Brief Title: Optical Frequency Domain Imaging (OFDI) and Vascular Healing After Stent Placement
Acronym: OFDI-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Henry A Liberman, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057208
Record Dates: First submitted 2012-11-07; First posted 2013-02-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty; Atherosclerosis; Wound Healing
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Non-diabetic patients receiving the Resolute stent (Experimental): Non-diabetic patients presenting with Acute Coronary Syndrome (ACS), receiving the Resolute stent.
  Interventions: Device: Resolute Integrity stent
- Diabetic patients receiving the Resolute stent (Experimental): Non-insulin dependent diabetes mellitus (NIDDM) patients presenting with Acute Coronary Syndrome (ACS), receiving the Resolute stent.
  Interventions: Device: Resolute Integrity stent

INTERVENTIONS:
Device: Resolute Integrity stent — Drug eluting stents used to treat coronary artery blockages

SUMMARY:
The use of drug eluting stents (DES) used to treat coronary artery blockages is limited by poor healing of the stented area. This will require the combined use of blood thinners such as aspirin and clopidogrel (i.e. dual anti-platelet therapy (DAPT)) to prevent complications such as clot formation on the stent which may lead to a heart attack. Diabetic patients and those presenting with a heart attack at the time of stent placement are at increased risk for clot formation. However, little is known of the healing responses after stent placement in these populations.

Currently all patients receiving DES are advised to complete DAPT for twelve months although more personalized durations of DAPT based on stent healing would reduce both clot formation and potential bleeding from the blood thinners, thereby improving the long-term safety of DES.

Intracoronary optical frequency domain imaging (OFDI) is a novel high resolution invasive imaging technique that has the ability to evaluate stent healing at follow-up. Among the commercially available coated stents used in the U.S., the zotarolimus eluting stents (RESOLUTE Integrity, Medtronic, Minneapolis, MN) has demonstrated superior healing in both preclinical and clinical studies.

The purpose of this trial is to determine the healing responses of the RESOLUTE Integrity stent as detected by OFDI in patients with and without diabetes presenting with ACS. Specifically, in this observational study, the study team will investigate non-insulin dependent diabetics and non-diabetics in the setting of ACS and RESOLUTE Integrity stent placement.

The investigators hypothesize that healing responses in patients with non-insulin dependent diabetes will be similar to those without diabetes presenting with ACS and that a majority of patients will demonstrate complete healing as determined by OFDI measurements.

DETAILED DESCRIPTION:
The long-term efficacy of drug eluting stents (DES) used to treat symptomatic coronary artery disease is limited by incomplete healing of the stented segment necessitating the use of dual anti-platelet therapy (DAPT) with aspirin and a thienopyridine to prevent these late thrombotic complications. Diabetic patients and those presenting with acute coronary syndrome (ACS) at the time of DES placement are at increased risk for late in stent thrombosis, however, little is known of the healing responses in these populations.

Currently all patients receiving DES are advised to complete DAPT for twelve months although more personalized durations of DAPT based on stent healing would reduce both thrombosis and bleeding, thereby improving the long-term safety of DES. Intracoronary optical frequency domain imaging (OFDI) is a novel high resolution invasive imaging modality with the potential to discern plaque morphology at stent placement and stent strut healing at follow-up. Among the commercially available coated stents used in the U.S., the zotarolimus eluting stents (RESOLUTE, Medtronic, Minneapolis, MN) has demonstrated superior endothelialization and long term safety data in both preclinical and clinical studies.

The purpose of this trial is to determine the healing responses to the RESOLUTE stent as detected by OFDI in patients with and without diabetes presenting with ACS. Specifically, investigators will 1) determine while using OFDI whether any difference in healing occurs in non-insulin dependent diabetic patients presenting with ACS after RESOLUTE stent placement at 6 months; 2) determine how initial plaque morphology and angiographic measures such as late loss correlate with stent strut healing; and 3) examine whether selected biomarkers have an utility in predicting stent strut healing by OFDI.

Investigators will conduct a clinical study that images subjects at baseline and at 6 months after stent placement with intracoronary OFDI. OFDI data will be utilized to determine plaque morphology prior to intervention, ensure adequate strut apposition and stent sizing immediately post deployment and to measure stent strut coverage at 6 month follow-up. Two follow-up imaging passes will be conducted to evaluate test-retest variability of the coverage measurement. In addition to assessing the feasibility of using the OFDI coverage metric in vivo, this data may provide information on the magnitude of coverage that can be expected at 6 months following RESOLUTE stents.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring percutaneous transluminal coronary interventions (PTCI) for acute coronary syndrome (ACS) and meeting criteria (as determined by the performing physician) for Resolute Integrity stent placement.

Exclusion Criteria:

* ST segment elevation MI (STEMI)
* stable angina
* current or planned pregnancy (for women of childbearing age)
* treatment of > 2 lesions during the index hospitalization
* insulin dependent diabetic patients at the time of stent placement
* use of overlapping stents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Liberman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JS, Jang IK, Fan C, Kim TH, Kim JS, Park SM, Choi EY, Lee SH, Ko YG, Choi D, Hong MK, Jang Y. Evaluation in 3 months duration of neointimal coverage after zotarolimus-eluting stent implantation by optical coherence tomography: the ENDEAVOR OCT trial. JACC Cardiovasc Interv. 2009 Dec;2(12):1240-7. doi: 10.1016/j.jcin.2009.10.006. PMID 20129551
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were selected from patients with acute coronary syndrome (ACS) presenting to Emory University Hospital Midtown for coronary angiography. Participants were recruited between September 2013 and September 2015.
Pre-assignment Details: Of the 24 individuals who signed the consent form, 16 were found to be ineligible to participate in the study, resulting in 8 participants who started the trial.
Groups:
- Non-diabetic Patients Receiving the Resolute Stent: Non-diabetic patients undergoing percutaneous transluminal coronary intervention (PTCI) for treatment of de novo native vessel coronary artery disease with the Resolute drug eluting stent
- NIDDM Patients Receiving the Resolute Stent: Non-insulin-dependent diabetes mellitus (NIDDM) patients undergoing percutaneous transluminal coronary intervention (PTCI) for treatment of de novo native vessel coronary artery disease with the Resolute drug eluting stent
Period: Overall Study
Arm/Group | Non-diabetic Patients Receiving the Resolute Stent | NIDDM Patients Receiving the Resolute Stent
Started | 7 | 1
6 Month Follow-up | 6 | 1
Completed | 6 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Individuals who consented to participate in the study and met all eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-diabetic Patients Receiving the Resolute Stent | NIDDM Patients Receiving the Resolute Stent | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Stent Coverage
Description: Assessment of vascular healing 6 months after Resolute Integrity placement in non-diabetic patients and patients with non-insulin dependent diabetes presenting with acute coronary syndrome (ACS) using optical frequency domain imaging (OFDI). Vascular healing will be measured by percent covered stents as determined by OFDI. A higher percentage of stent coverage indicates increased endothelial regrowth, which is an essential component for the maintenance of long-term luminal patency.
Time Frame: 6 months
Population: Participants included in the analyses for this outcome are those who completed the 6 month follow-up imaging to assess vascular healing. Optical frequency domain imaging (OFDI) was not performed on two participants in the non-diabetic study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-diabetic Patients Receiving the Resolute Stent | NIDDM Patients Receiving the Resolute Stent
Number analyzed (Participants) | 5 | 1
Participants
  85% up to 90% stent coverage | 1 | 0
  90% up to 95% stent coverage | 3 | 1
  95% or greater percent stent coverage | 1 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events for 6 months after having the study procedure. Adverse events were followed until the event subsided or, in the case of permanent impairment, the event stabilized and the overall clinical outcome was ascertained.
Description: Participants were instructed to notify the research physician of any adverse effects of treatment, including those that are anticipated with this treatment.
Arm/Group | Non-diabetic Patients Receiving the Resolute Stent | NIDDM Patients Receiving the Resolute Stent
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/1
Other Adverse Events (participants affected / at risk) | 2/7 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-diabetic Patients Receiving the Resolute Stent (N=7) | NIDDM Patients Receiving the Resolute Stent (N=1)
Heart attack symptoms (Cardiac disorders) | 1 (1) | 0 (0) — Lethargy, back pain, chest pain, panic attack resulted in a repeat angiogram. The Left Anterior Descending (LAD) artery sent was patent and the symptoms resolved without treatment.
Coronary occlusion (Vascular disorders) | 1 (1) | 0 (0)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0)
Iliac occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-diabetic Patients Receiving the Resolute Stent (N=7) | NIDDM Patients Receiving the Resolute Stent (N=1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Elevated creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to low enrollment there were not enough participants to provide 80% power for the comparison between the study arms, therefore, statistical analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes